CLINICAL TRIAL: NCT04920604
Title: Anesthetic and Perioperative Risk Assessment Before Programmed Surgery: Anesthetic Teleconsultation Versus Face-to-face Anesthesia Consultation.
Acronym: TELANESTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NIMAO/2020-2/EM-01; 2021-A00311-40 (Other: ANSM)
Record Dates: First submitted 2021-05-27; First posted 2021-06-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Telemedicine; Anesthesia; Consultation, Remote

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teleconsultation (Experimental)
  Interventions: Other: Remote anesthesia consultation
- Control group (Active Comparator)
  Interventions: Other: Face-to-face anesthesia consultation

INTERVENTIONS:
Other: Face-to-face anesthesia consultation — The anesthesia consultation is carried out in person in accordance with the usual management.
  Arms: Control group
Other: Remote anesthesia consultation — Anesthesia consultation is carried out in teleconsultation via the "Téléo" web application (audio and video) at the patient's home on a computer or smartphone. This application allows sending and receiving documents identical to those during the face-to-face consultation.
  Arms: Teleconsultation

SUMMARY:
The anesthesia safety decree made it compulsory in 1994 to carry out a pre-anesthesia consultation before any operative or interventional act. With the inclusion of telemedicine in the Public Health Code then the publication of Addendum 6 in 2018 and finally the derogatory decree in March 2020, it is possible to perform and bill for pre-anesthesia consultation via telemedicine.

The consultation is always followed by a pre-anesthetic visit upon admission of the patient the day before or the day of the operation to verify the information recorded during the consultation and the patient's state of health. This identifies elements omitted during the pre-anesthesia consultation (face-to-face or remotely) and reduces the risks of potential postponement.

The study investigators hypothesize that there would be no difference in the quality of the information given, the collection of medical, paramedical and medication elements and the evaluation of the operative risk in anesthesia consultation via teleconsultation versus face-to-face. The critical points are the medication reconciliation of the patient's treatments, the overall assessment of the operative risk and anticipated difficulty of access to the airways (mouth opening: ≥ or <35 mmm).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient with scheduled surgical intervention (outpatient or hospitalization) at the Nîmes University Hospital requiring a preoperative anesthesia consultation.
* Patient with computer equipment at home allowing the use of the Téléo software (computer equipment with web cam, audio and microphone or smartphone).

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient who has already had an anesthesia consultation for surgery within the previous 6 months.
* Emergency or radiology and / or interventional surgery (eg. gastroscopy, biopsy under scanner, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Elevated American Society of Anesthesiologists (ASA) score in each group | anesthesia consultation = 1 week to 3 months after inclusion
  Yes/no for if score=3-4
Elevated American Society of Anesthesiologists (ASA) score in each group | pre-anesthetic visit = 9 days to 3 months+7 days after inclusion
  Yes/no for if score=3-4
Difficulty in accessing airways each group | anesthesia consultation = 1 week to 3 months after inclusion
  Yes/no for mouth opening ≥35 mm
Difficulty in accessing airways each group | pre-anesthetic visit = 9 days to 3 months+7 days after inclusion
  Yes/no for mouth opening ≥35 mm
Medication conciliation performed during the anesthesia consultation each group | pre-anesthetic visit = 9 days to 3 months+7 days after inclusion
  Yes/no: adaptations of selected therapies: anticoagulants, anti-aggregants, anti-hypertension, antidiabetics
Medication conciliation performed during the anesthesia consultation each group | anesthesia consultation = 1 week to 3 months after inclusion
  Yes/no: adaptations of selected therapies: anticoagulants, anti-aggregants, anti-hypertension, antidiabetics
Difference between groups in composite score of above outcomes (elevated ASA score, difficulty accessing airways and medication conciliation) | pre-anesthetic visit = 9 days to 3 months+7 days after inclusion
  Difference in number of yes/no answers at anesthesia consultation compared to pre- anesthetic visit
Difference between groups in composite score of above outcomes (elevated ASA score, difficulty accessing airways and medication conciliation) | anesthesia consultation = 1 week to 3 months after inclusion
  Difference in number of yes/no answers at anesthesia consultation compared to pre- anesthetic visit

SECONDARY OUTCOMES:
Number of canceled surgeries in each group | Day 2 after pre-anesthetic visit
  Yes/no surgery not performed on the scheduled day and / or postponed > 2 days
Reason for cancellation of surgery | Day 2 after pre-anesthetic visit
  Description noted in electronic clinical report form
Number of delayed surgeries in each group | Day 2 after pre-anesthetic visit
  Yes/no surgery not performed on the scheduled day and / or postponed ≤ 2 days
Reason for delayed surgery | Day 2 after pre-anesthetic visit
  Description noted in electronic clinical report form
Complication rate in perioperative and immediate postoperative period | 2 days post-operatively
  % patients with a complication
Rate of anesthesia consultation rescheduling in each group | 2 days after pre-anesthetic visit
  Number of consultations rescheduled
Reason for rescheduling | 2 days after pre-anesthetic visit
  Description noted in electronic clinical report form
Global patient satisfaction | pre-anesthetic visit = 9 days to 3 months+7 days after inclusion
  satisfaction on a visual analog scale 0-10
Satisfaction on the delivery of the information | pre-anesthetic visit = 9 days to 3 months+7 days after inclusion
  6-item custom questionnaire completed on a Likert 0 - 5 scale for all patients plus 6 questions specific for control group and 7 for intervention group
Ecological impact of the consultation in each group | pre-anesthetic visit = 9 days to 3 months+7 days after inclusion
  Carbon impact (CO2 generated) of number of km between the patient's home and the hospital
Economic impact of the consultation in each group | pre-anesthetic visit = 9 days to 3 months+7 days after inclusion
  Cost in euros of cost of travel and time at work missed
Rate of presence of the usual treatment prescription | During the anesthesia consultation = 1 week to 3 months after inclusion
  Yes/no
Rate of presence of the completed health questionnaire | During the anesthesia consultation = 1 week to 3 months after inclusion
  Yes/no
Rate of presence of specialist consultation reports less than 1 year old | During the anesthesia consultation = 1 week to 3 months after inclusion
  Yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Estelle Morau, Principal Investigator — CHU Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France

REFERENCES:
- [Result] Morau E, Blanc A, Boisson C, Sawyers T, Lefrant J, Cuvillon P. Telemedicine for Preanesthesia Consultations During the First COVID-19 Lockdown. Telemed J E Health. 2023 Apr;29(4):621-624. doi: 10.1089/tmj.2022.0143. Epub 2022 Jul 26. PMID 35877785